CLINICAL TRIAL: NCT06988670
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Trial Investigating the Safety, Tolerability and Efficacy of EXT608 in Adults With Hypoparathyroidism
Brief Title: A Phase 2 Trial Investigating the Safety, Tolerability and Efficacy of EXT608 in Adults With Hypoparathyroidism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Extend Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EXT608-201; R01FD007824 (FDA); R44DK138647 (NIH)
Record Dates: First submitted 2025-04-30; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hypoparathyroidism
Keywords: hypopara
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): EXT608 solution for injection, administered subcutaneously once-weekly, with multiple ascending doses (MAD) with a starting dose of 50 ug for 4 weeks, continuing to individualized dosing for 8 weeks
  Interventions: Drug: EXT608
- Placebo (Placebo Comparator): Placebo solution, administered subcutaneously once-weekly, with multiple ascending doses (MAD) with a fixed dose for 4 weeks, continuing to variable dosing for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EXT608 — Modified version of parathyroid hormone attached to vitamin D to extend half-life
  Arms: Active
Other: Placebo — Placebo for injection
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety, tolerability and efficacy of EXT608 in adults with hypoparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to personally provide written, signed, and dated informed consent to participate in the study.
2. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
3. Male or female between 18 and 65 years of age. Male participants with female partners of child bearing potential must agree to use barrier contraception, e.g., condoms plus spermicide, from administration of the study drug until at least 3 months after administration of the study drug. Abstinence from heterosexual intercourse from administration of study drug until at least 3 months after administration of study drug is acceptable if it is in accordance with the participant's lifestyle. Female participants should be either surgically sterile (had a bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy, or hysterectomy), postmenopausal (defined as 12 months with no menses prior to screening and a serum follicle stimulating hormone in the postmenopausal range at screening), or, if of child bearing potential, must be non-lactating and willing to use a highly effective method of birth control for 30 days prior to administration of study drug and agree to continued use of this method until at least 3 months after administration of study drug.
4. Participants have a history of hypoparathyroidism for 12 months at least, with PTH levels below the LLN with concomitant serum calcium < 9 mg/dL.
5. Participants are treated with a daily dose > 750 mg elemental calcium if using > 0.25 µg/day calcitriol, or a daily dose > 1000 mg elemental calcium if not using calcitriol.
6. Participants have normal blood levels of 25-hydroxyvitamin D (i.e. > 20 ng/dL or > 75 nmol/L) and not above 1.5 times the upper limit of normal.
7. Participants have normal thyroid test results for 3 months at least while taking a stable dose of thyroid medication or no medication.
8. Participants have a BMI < 35 kg/m2.
9. Albumin-adjusted serum calcium level should be between the lower half and the middle of the normal range upon randomization into the study.

Exclusion Criteria:

1. Participants with hypoparathyroidism due to an activating mutation of the calcium sensing receptor, pseudohypoparathyroidism, any non-hypoparathyroidism disease that may affect calcium metabolism or phosphor-calcium homeostasis, or requiring parenteral calcium infusions.
2. Unwillingness to use a diary deployed on a smartphone daily for recording vitamin D, active vitamin D, calcium, magnesium and study drug doses as well as periodic symptom reporting.
3. Participants with a history of neoplasia (except thyroid cancer) with no sign of recurrence 5 years after diagnosis.
4. Participants with a history of or active GI tract disease that may impact the absorption of calcium (e.g. malabsorption).
5. Participants with a history of severe hypocalcemia leading to seizures or cardiac arrhythmias within 6 months prior to screening.
6. Participants with chronic kidney disease (eGFR < 30 ml/min) or active nephrolithiasis (needing pain medication in the last 6 months).
7. Participants taking the following medications within the respective exclusion period:

   * Proton pump inhibitors (4 weeks)
   * Bisphosphonates (3 months)
   * Parathyroid hormone, PTH analogs (6 months)
   * Thiazide diuretics (14 days)
   * Calcitonin or calcinet hydrochloride (3 months)
8. Participant has increased CV proarrhythmic potential:

   1. Participant has a QT interval with Fridericia's correction method (QTcF) >450 ms or PR outside the range of 120 to 220 ms, confirmed with one repeat testing, at the Screening Visit or Inpatient Check-in (Day -1) Visit.
   2. A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
   3. The use of concomitant medications that prolong the QT/QTc interval.
9. Chronic/severe cardiac disease including, but not limited to, cardiac insufficiency, unstable angina, arrhythmias, bradycardia (resting heart rate <60 beats/minute), or hypotension (systolic and diastolic blood pressures <100 and 60 mmHg, respectively).
10. Any condition or disease that, in the opinion of the investigator, may interfere with a participant's participation or may confound the interpretation of safety or efficacy in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of multiple subcutaneous (SC) escalating dose levels of EXT608 in participants with hypoparathyroidism by determining frequency and severity of treatment emergent adverse events and post-dose change in lab results | From enrollment until the end of treatment at 12 weeks
  Frequency and severity of treatment emergent adverse events; frequency and severity of post-dose change from baseline in laboratory analyses; percentage of participants with injection site reactions

SECONDARY OUTCOMES:
Assess the pharmacokinetics (PK) of multiple SC doses of EXT608 given over 4 weeks in participants with hypoparathyroidism by determining Area Under the Curve (AUC) | From enrollment until 4 weeks
  Determine Area Under the Curve (AUC)
Assess the pharmacokinetics (PK) of multiple SC doses of EXT608 given over 4 weeks in participants with hypoparathyroidism by determining drug half-life | From enrollment until 4 weeks
  Determine drug half-life
Assess the clinical efficacy of multiple fixed SC doses of EXT608 given over 4 weeks (at week 4), and individualized dosing after an additional 8 weeks (at week 12) in participants with hypoparathyroidism by assessing serum calcium | From enrollment until the end of treatment at 12 weeks
  Proportion of participants with normal serum calcium
Assess the clinical efficacy of multiple fixed SC doses of EXT608 given over 4 weeks (at week 4), and individualized dosing after an additional 8 weeks (at week 12) in participants with hypoparathyroidism by assessing supplementation | From enrollment until the end of treatment at 12 weeks
  Assess change from baseline of daily ingested amount of oral calcium, vitamin D supplements

CONTACTS AND LOCATIONS:
Locations (1):
- Trial Site, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided
Will be determined upon completion of the study.